CLINICAL TRIAL: NCT03150940
Title: Changing the Pulse of Athletics: Applying a Standardized Cardiac Athletic Screening for NCAA Athletes
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00069459
Record Dates: First submitted 2016-04-14; First posted 2017-05-12 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Athletes Heart
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duke University Athletes: Division 1 Athletes, participating in obligatory screening prior to athletic competition every summer. The investigators are observing required study outcomes (ECGs, history and physicals, and ultrasounds) to see what is useful in the screening.
  * ECG: 12 lead electrocardiogram that visualizes cardiac activity
  * history and physical: background information about athlete's and their family history
  * ultrasound: bedside cardiac ultrasound to visualize 2D imaging of structural cardiac function
  Interventions: Diagnostic Test: ECG; Diagnostic Test: bedside cardiac ultrasound

INTERVENTIONS:
Diagnostic Test: ECG — 12 lead electrocardiogram used to demonstrate cardiac function
Diagnostic Test: bedside cardiac ultrasound — bedside cardiac ultrasound to see 2D images of each participants heart. Without the use of radiation.

SUMMARY:
This is a study supported by Duke Sports Cardiology and Duke Sports Medicine with the intent to enhance the cardiovascular screening of collegiate athletes from a regional to nationally recognized program to understand and eventually reduce cardiovascular events in athletes. The data from this ongoing registry will be used to better understand, refine, and improve the current cardiovascular Duke Athlete Screening process and use this experience as a role model to expand across the ACC.

DETAILED DESCRIPTION:
The purpose of this study is to screen for and determine the prevalence of structural, functional, or electrophysiologic cardiac abnormalities in a population of young athletes using bedside cardiac ultrasound, electrocardiogram (ECG) and a physical exam.

The investigators will attempt to answer the question regarding the feasibility of screening all collegiate athletes with bedside cardiac ultrasound, ECG, and history/physical exams results in a higher sensitivity for abnormalities than screening using ECG and physical exams alone. The investigators will also analyze the cost and cost effectiveness of screening the young athlete population with bedside cardiac ultrasound. Costs will be calculated to include the amount of dollars spent on equipment, gels, and other supplies, but will not include the cost of performing the bedside cardiac ultrasound, which will be assumed as part of the physical exam. Additionally, the investigators will be gathering a number of data markers from the bedside cardiac ultrasound, including but not limited to right ventricular and left ventricular cavitary size, septal wall thickness, free ventricle wall on RV, and free ventricle wall on LV, in evaluation of the athlete's heart. The importance of these measurements is for the continued knowledge and data set analysis collection as there is limited known athletic cardiac measurements. There is minimal risk involved in this study. The investigators believe that by adding bedside cardiac ultrasound to the history, physical, and ECG, it will increase the sensitivity and specificity of screening for these life-threatening abnormalities in young athletes, and reduce the morbidity and mortality associated with these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Athletes with previous known cardiac abnormality will be included in the study. Participants in the cardiovascular screening are young student athletes of Duke University between the ages of 18-22, of both sexes participating in their respective athletic pre-participation physical examination. Anyone who participates in NCAA Division 1 collegiate athletics is eligible to participate in the study.

Exclusion Criteria:

* Exclusions to this study include any walk-on athletes, or those not deemed a part of Duke Athletics prior to the commencement of the academic year. Also excluded will be anyone less than 18 years of age. Student athletes who do not agree to the study consent will be excluded.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in NCAA Division 1 collegiate athletics at Duke University are eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Estimates of false positive rates for use of ultrasound and electrocardiogram | 1 month
  Comparing the false positive rates of use of ultrasound and electrocardiogram

SECONDARY OUTCOMES:
To compare the rate of accuracy for athletic screenings. | 1 month
  To compare how observing data collectors make assessments for collected data.

OTHER OUTCOMES:
The feasibility of quality data collection. | 1 month
  As measured by estimated cost and access to resources.
The mean estimated time to complete this study | 1 month
  Measured by work hours and time to collect the data

CONTACTS AND LOCATIONS:
Overall Officials: Blake Boggess, DO, Principal Investigator — Associate Professor of Clinical Sports Medicine
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maron BJ, Haas TS, Murphy CJ, Ahluwalia A, Rutten-Ramos S. Incidence and causes of sudden death in U.S. college athletes. J Am Coll Cardiol. 2014 Apr 29;63(16):1636-43. doi: 10.1016/j.jacc.2014.01.041. Epub 2014 Feb 26. PMID 24583295
- [Background] Maron BJ, Doerer JJ, Haas TS, Tierney DM, Mueller FO. Sudden deaths in young competitive athletes: analysis of 1866 deaths in the United States, 1980-2006. Circulation. 2009 Mar 3;119(8):1085-92. doi: 10.1161/CIRCULATIONAHA.108.804617. Epub 2009 Feb 16. PMID 19221222
- [Background] Sheikh N, Papadakis M, Ghani S, Zaidi A, Gati S, Adami PE, Carre F, Schnell F, Wilson M, Avila P, McKenna W, Sharma S. Comparison of electrocardiographic criteria for the detection of cardiac abnormalities in elite black and white athletes. Circulation. 2014 Apr 22;129(16):1637-49. doi: 10.1161/CIRCULATIONAHA.113.006179. Epub 2014 Mar 11. PMID 24619464
- [Background] Maron BJ, Pelliccia A. The heart of trained athletes: cardiac remodeling and the risks of sports, including sudden death. Circulation. 2006 Oct 10;114(15):1633-44. doi: 10.1161/CIRCULATIONAHA.106.613562. No abstract available. PMID 17030703